CLINICAL TRIAL: NCT05890599
Title: Randomized Multicenter Clinical Trial: Yoga Versus Health Education for the Treatment of Persistent Fatigue in Patients With Post COVID-19 Syndrome
Brief Title: Yoga Versus Health Education for the Treatment of Persistent Fatigue in Patients With Post COVID-19 Syndrome
Acronym: YoFaPoCo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S00766-RBK
Record Dates: First submitted 2023-06-02; First posted 2023-06-06 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Post-COVID-19 Syndrome; Fatigue Post Viral
Keywords: Fatigue; Covid
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yoga Therapy (Experimental): 12 week yoga program, one weekly session of 90 minutes each, plus 2 times weekly 30 minutes of self practice.
  Interventions: Behavioral: Yoga Therapy
- Health Education (Active Comparator): 12 week health education program, one weekly session of 90 minutes each, plus 2 times weekly 30 minutes of self practice.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Yoga Therapy — The range of interventions is based on previous studies on yoga interventions specifically for fatigue patients as well as on recommendations, for example, from the WHO. The yoga therapy includes 3 elements: yoga postures (asanas), breathing techniques (pranayama) and relaxation moments.
  Emphasis on postures and breathing techniques that are considered to be effective for fatigue symptoms, as well as specific breathing exercises to strengthen the respiratory muscles and increase lung volume.
  Arms: Yoga Therapy
Behavioral: Health Education — Health education courses are conducted on-site once a week for 90 minutes over a 12-week period by a psychologist with clinical experience. The courses are didactic in nature and consist of lectures on topics of interest to patients with post-COVID syndrome and fatigue, followed by questions and discussion sessions. Topics include information on post-COVID syndrome and fatigue, an introduction to self-help for post-viral symptoms, psychosocial problems and fatigue, relaxation and stress management, nutrition, sleep hygiene, exercise, respecting one's own limits, acceptance, finding meaning, and achieving goals.
  Arms: Health Education

SUMMARY:
Evaluation of the short- and medium-term effect of a yoga intervention in addition to routine care compared to health education in addition to routine care on fatigue in patients with post covid syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 diagnosis
* Follow-up symptoms of ≥ 12 weeks
* Persistent fatigue (scores ≥4 on the binomial Chalder Fatigue Scale).
* Self-assessment that fatigue was a consequence of COVID-19 disease
* Age 18-65 years

Exclusion Criteria:

* Chronic medical conditions or regular use of medications associated with fatigue
* Indication of health cause of fatigue other than post-COVID.
* Indication of other factors as the main cause of fatigue
* Physical limitations that do not allow participation in the yoga intervention
* Pregnancy, breastfeeding
* Concurrent participation in other clinical trials
* Current yoga practice

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Fatigue | 12 weeks
  The chalder fatigue scale is used to assess the severity of fatigue within the last 4 weeks. It contains 11 questions in a four-step answer format (0-4), 7 of which refer to the degree of physical fatigue and 4 to the degree of mental fatigue. In its binomial evaluation (range 0-11) it can be used with a cut-off of (≥ 4) to divide patients into those with and those without fatigue.

SECONDARY OUTCOMES:
Fatigue | 24 weeks
  The chalder fatigue scale is used to assess the severity of fatigue within the last 4 weeks. It contains 11 questions in a four-step answer format (0-4), 7 of which refer to the degree of physical fatigue and 4 to the degree of mental fatigue. In its binomial evaluation (range 0-11) it can be used with a cut-off of (≥ 4) to divide patients into those with and those without fatigue.
Health related quality of life SF-12 | 12 weeks
  Short Form 12 Health Survey Questionnaire, The SF-12 represents the most commonly used instrument in clinical trials to assess generic quality of life. The questionnaire captures 8 different subscales, which are combined into a physical and a psychological summated scale.
Health related quality of life SF-12 | 24 weeks
  Short Form 12 Health Survey Questionnaire, The SF-12 represents the most commonly used instrument in clinical trials to assess generic quality of life. The questionnaire captures 8 different subscales, which are combined into a physical and a psychological summated scale.
Health related quality of life EQ-5D-5L | 12 weeks
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. In this study, the EQ-5D-5L is used for cost-effectiveness analysis, together with healthcare-related costs.
Health related quality of life EQ-5D-5L | 24 weeks
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. In this study, the EQ-5D-5L is used for cost-effectiveness analysis, together with healthcare-related costs.
Psychological symptoms | 12 weeks
  The Hospital Anxiety and Depression Scale asks 14 questions, of which 7 are about anxiety and 7 about depression in patients with physical illnesses and physical complaints. More precisely, it measures the self-assessed severity of patients' anxious and depressive symptoms in relation to the past week.
Psychological symptoms | 24 weeks
  The Hospital Anxiety and Depression Scale asks 14 questions, of which 7 are about anxiety and 7 about depression in patients with physical illnesses and physical complaints. More precisely, it measures the self-assessed severity of patients' anxious and depressive symptoms in relation to the past week.
Sleep quality | 12 weeks
  The Pittsburgh Sleep Quality Index (PSQI) assesses the quality of sleep over the past 4 weeks using 24 questions, 17 for self-assessment and 7 for external assessment. It is used clinically to monitor patients with sleep disorders and to screen for sleep disorders in epidemiological studies. In this study, only the 17 self-assessment items are collected.
Sleep quality | 24 weeks
  The Pittsburgh Sleep Quality Index (PSQI) assesses the quality of sleep over the past 4 weeks using 24 questions, 17 for self-assessment and 7 for external assessment. It is used clinically to monitor patients with sleep disorders and to screen for sleep disorders in epidemiological studies. In this study, only the 17 self-assessment items are collected.
Stress | 12 weeks
  The current stress perception of the patients is assessed by means of the Perceived Stress Scale (PSS-10). This measures the current subjective perceived stress of the patients on the basis of 10 items.
Stress | 24 weeks
  The current stress perception of the patients is assessed by means of the Perceived Stress Scale (PSS-10). This measures the current subjective perceived stress of the patients on the basis of 10 items.
Post-exertional malaise | 12 weeks
  Post-exertional malaise (PEM) is a delayed worsening of symptoms that occurs after minimal physical or mental activity. The DePaul-Symptom Questionaire (DSQ) is used to asses PEM.
Post-exertional malaise | 24 weeks
  Post-exertional malaise (PEM) is a delayed worsening of symptoms that occurs after minimal physical or mental activity. The DePaul-Symptom Questionaire (DSQ) is used to asses PEM.
Body awareness | 12 weeks
  The Body Awareness Questionnaire (BAQ) assesses participants' subjective body awareness in four subdimensions: note responses or changes in body processes, predict bodily reaction, sleep-wake cycle, and onset of illness. The validated single-factor German version consists of 17 questions on a 7-point Likert scale from 1 (not at all true about me) to 7 (very true about me). The values of the individual items are added together to form a total score. Body awareness will be used in mediation analyses of treatment effects.
Body awareness | 24 weeks
  The Body Awareness Questionnaire (BAQ) assesses participants' subjective body awareness in four subdimensions: note responses or changes in body processes, predict bodily reaction, sleep-wake cycle, and onset of illness. The validated single-factor German version consists of 17 questions on a 7-point Likert scale from 1 (not at all true about me) to 7 (very true about me). The values of the individual items are added together to form a total score. Body awareness will be used in mediation analyses of treatment effects.
Self-Efficacy | 12 weeks
  The Arthritis Self-Efficacy Scale (ASES) was originally developed in 1989 as part of the Stanford Arthritis Self-Management Study to assess self-efficacy in arthritis patients and has since been used to assess it in many disease conditions. A short version (ASES-8/ASES-D) has been validated. This version surveys in scale level 1-10 the perceived ability to deal with occurring symptoms such as: Pain or fatigue. Self-efficacy will be used in mediation analyses of treatment effects.
Self-Efficacy | 24 weeks
  The Arthritis Self-Efficacy Scale (ASES) was originally developed in 1989 as part of the Stanford Arthritis Self-Management Study to assess self-efficacy in arthritis patients and has since been used to assess it in many disease conditions. A short version (ASES-8/ASES-D) has been validated. This version surveys in scale level 1-10 the perceived ability to deal with occurring symptoms such as: Pain or fatigue. Self-efficacy will be used in mediation analyses of treatment effects.
Adverse events | Week 0, 1-12, 13 and 25
  Adverse events and serious adverse events are documented. Adverse events include any adverse symptoms, illnesses, disorders, or accidents that occur during the course of the study. Serious adverse events include events occurring during the course of the study that are immediately life-threatening and/or result in serious health problems (specifically, requiring unanticipated hospitalization or prolongation of hospitalization, or resulting in serious disability or incapacitation). Adverse events (including PEM) and serious adverse events will be documented by participants on a weekly basis throughout the intervention period. Participants will be instructed to immediately notify the study site upon the occurrence of any serious adverse event. The severity as well as the possible causal relationship with the intervention will be assessed by the study physician.
C-reactive proteine | 12 weeks
  CRP as marker of pro-inflammatory cytokine activity, from blood samples.
C-reactive proteine | 24 weeks
  CRP as marker of pro-inflammatory cytokine activity, from blood samples.
Interleukine-6 | 12 weeks
  IL-6, as marker of pro-inflammatory cytokine activity, from blood samples.
Interleukine-6 | 24 weeks
  IL-6, as marker of pro-inflammatory cytokine activity, from blood samples.
D-dimer | 12 weeks
  D-dimer, as a by-product of the blood clotting and break-down process that can be measured via analysis of a blood sample
D-dimer | 24 weeks
  D-dimer, as a by-product of the blood clotting and break-down process that can be measured via analysis of a blood sample
Lactate dehydrogenase | 12 weeks
  Lactate dehydrogenase (LDH), measuring the amount of LDH in the blood. Lactate dehydrogenase is an enzyme that the body uses during the process of turning sugar into energy for your cells to use.
Lactate dehydrogenase | 24 weeks
  Lactate dehydrogenase (LDH), measuring the amount of LDH in the blood. Lactate dehydrogenase is an enzyme that the body uses during the process of turning sugar into energy for your cells to use.
Leukocytes and lymphocytes | 12 weeks
  Leukocytes and lymphocytes, from blood samples.
Leukocytes and lymphocytes | 24 weeks
  Leukocytes and lymphocytes, from blood samples.
Hand grip strength | 12 weeks
  Repeated measurement of hand strength can help detect physical decline and inflammatory processes Hand grip strength measurement can be an invaluable tool for monitoring physical performance decline.
Hand grip strength | 24 weeks
  Repeated measurement of hand grip strength can help detect physical decline and inflammatory processes Hand strength measurement can be an invaluable tool for monitoring physical performance decline.
Movement tracking | 12 weeks
  General tracking of patients' movement habits via activity monitor
Movement tracking | 24 weeks
  General tracking of patients' movement habits via activity monitor
Heart rate variability | 12 weeks
  24-hour measurement of heart rate variability (HRV) to determine the functionality of the participant's autonomic nervous system. A 3-channel ECG recorder (SRA/Multi-ECG recorder, SR-Medizinelektronik, Stuttgart, Germany) is used. Several HRV time-domain and HRV frequency-domain measures will be evaluated and analyzed for the total day and night (sleeping time) period as well as for 5-minutes-intervals within these two periods (SDNN, RMSSD, pNN50, SDANN, SDNNI, VLF power, LF power, HF power, LF/HF).
Heart rate variability | 24 weeks
  24-hour measurement of heart rate variability (HRV) to determine the functionality of the participant's autonomic nervous system. A 3-channel ECG recorder (SRA/Multi-ECG recorder, SR-Medizinelektronik, Stuttgart, Germany) is used. Several HRV time-domain and HRV frequency-domain measures will be evaluated and analyzed for the total day and night (sleeping time) period as well as for 5-minutes-intervals within these two periods (SDNN, RMSSD, pNN50, SDANN, SDNNI, VLF power, LF power, HF power, LF/HF).
Cost for Patient Questionnaire (CoPaQ) | 12 weeks, 24 weeks
  Direct medical and non-medical costs are collected using this questionnaire. The questionnaire is a modified version of the Cost for Patient Questionnaire (CoPaQ), designed to collect all information on health care costs.

OTHER OUTCOMES:
Therapy rationale and therapy expectancy | Week 0
  The Credibility Expectancy Questionnaire (CEQ) published by Ametrano, et al. 2011 and validated as German version by Rieke, et al. 2013 is used to measure Therapierationale and Therapieerwartung at baseline. It measures these over 6 items using 9-point Likert scales.
Personality dimensions | Week 0
  Big-Five-Inventory-10 (BFI-10) is used to assess personality dimensions based on the big-5 model.
Qualitative Interviews | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Holger Cramer, Professor, Study Director — University Hospital Tübingen
Locations (1):
- Bosch-Health-Campus, Stuttgart, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cramer H, Morchen L, Vagedes J, Klenk J, Jager S, Schleinzer A, Anheyer D, Bilc M, Schroter M, Kessler C, Jeitler M. Yoga versus health education for persistent fatigue in patients with post-COVID-19 syndrome: protocol for a multicentre randomised controlled trial. BMJ Open. 2025 Oct 23;15(10):e107840. doi: 10.1136/bmjopen-2025-107840. PMID 41130694